CLINICAL TRIAL: NCT00042588
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Safety and Efficacy Study of Hospitalized Patients With Community-Acquired Pneumonia and Sepsis
Brief Title: A Safety and Efficacy Study of Hospitalized Patients With Community-Acquired Pneumonia and Sepsis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ICOS Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPN01; EPN01
Record Dates: First submitted 2002-08-01; First posted 2002-08-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-01

CONDITIONS: Pneumonia; Sepsis
Keywords: Safety and Efficacy; Community-Acquired Pneumonia, Sepsis
MeSH Terms: conditions — Pneumonia; Sepsis; Community-Acquired Pneumonia

INTERVENTIONS:
Drug: Recombinant Chimeric Monoclonal Antibody

SUMMARY:
The objective of this study is to demonstrate the safety and efficacy of IC14 in the treatment of hospitalized patients with community-acquired pneumonia and sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of community-acquired pneumonia.
* Evidence of systemic inflammatory response to infection.

Exclusion Criteria:

* Atypical or viral pneumonia based on clinical or epidemiologic suspicion by the investigator.
* Presence of organ failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-05

CONTACTS AND LOCATIONS:
Locations (1):
- ICOS Corporation, Bothell, Washington, United States